CLINICAL TRIAL: NCT03559387
Title: A Randomized and Open-label Dose-finding, Ph. 2, Efficacy, Safety, and Pharmacokinetic Study of Once-per-cycle Prophylactic Injections of ANF-RHO™ Versus Pegfilgrastim (Neulasta®) in Non-metastatic Breast Cancer Patients at High-risk of Chemotherapy-induced Neutropenia
Brief Title: Randomized Phase 2, Dose-finding Efficacy, Safety Study of ANF-RHO™ Versus Neulasta® in Chemotherapy-Induced Neutropenia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study redesign
Sponsor: Prolong Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PGFN-001
Record Dates: First submitted 2018-05-10; First posted 2018-06-18 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2018-06

CONDITIONS: Chemotherapy-induced Neutropenia
MeSH Terms: interventions — pegylated granulocyte colony-stimulating factor; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ANF-RHO™ (Experimental): Subjects will receive the ANF-RHO™ dose with a volume equivalent to 10 µg/kg, 20 µg/kg and 30 µg/kg as a subcutaneous injection.
  Interventions: Drug: ANF-RHO™
- Neulasta® (Active Comparator): Neulasta® will be administered to the subjects at a dose of 6.0 mg in 0.6 ml as a subcutaneous injection.
  Interventions: Drug: Neulasta®

INTERVENTIONS:
Drug: ANF-RHO™ — Subjects randomized to the ANF-RHO™ treatment arm will receive the investigational product on Day 1(day of chemotherapy treatment) of each Chemotherapy cycle. ANF-RHO™ will be administered to the subjects as a subcutaneous injection. Subjects will receive the ANF-RHO™ dose with a volume equivalent to 10 µg/kg, 20 µg/kg and 30 µg/kg.
  ANF-RHO™ is provided as a single-use glass vial containing 1.0 ml of solution at a concentration of 5 mg/ml
  Other Names: Pegylated Granulocyte Colony-Stimulating Factor (PEG-GCSF)
  Arms: ANF-RHO™
Drug: Neulasta® — Subjects randomized to the Neulasta® treatment arm will receive the comparator drug on Day 2(day after chemotherapy treatment) of each Chemotherapy cycle. Neulasta® will be administered to the subjects at a standard dose of 6.0 mg in 0.6 ml as a subcutaneous injection.
  Neulasta® is also provided as a single-use pre-filled syringe.
  Other Names: Pegylated Granulocyte Colony-Stimulating Factor (PEG-GCSF)
  Arms: Neulasta®

SUMMARY:
Randomized, Open-Label study to determine the dose, efficacy, safety and pharmacokinetic profile of ANF-RHO™ with once-per-cycle injection in comparison with Neulasta in Breast Cancer patients at high risk of developing Chemotherapy-Induced Neutropenia

DETAILED DESCRIPTION:
Forty Eight (48) adult female, chemotherapy treatment-naïve, stage I to III, breast cancer patients scheduled to receive FEC100 (3 cycles)/docetaxel (3 cycles) myelosuppressive chemotherapy will be enrolled into the study after they meet all the inclusion/exclusion criteria. Four (4) Cohorts of 12 patients each will be studied; they will be randomized either in the ANF-RHO™ treatment arm at different doses (10 μg/kg, 20 μg/kg, or 30 μg/kg, for the cohorts 1-3, respectively) or Neulasta® (6 mg / 0.6 ml SC injection, for cohort 4). For the cohorts 1-3, 12 patients from each of the respective ANF-RHO™ cohorts will be randomized with four patients from cohort 4 (Neulasta®). Patients in the ANF-RHO™ cohorts will receive study drug on Day 1 of each Chemotherapy cycle. Patients in the Neulasta® cohort will receive study drug on Day 2 of each Chemotherapy cycle. Doses of ANF-RHO™/Neulasta® will be provided for a total of 6 cycles (21 days each). The total duration of the study 129 ± 2 days (126 Days of treatment period followed by end of study visit)

ELIGIBILITY:
Inclusion Criteria:

1. Adult female patients, 18 years of age or older
2. Signed and dated written consent/assent by the patient or legally authorized representative
3. Histologically confirmed non-metastatic breast cancer
4. ECOG performance status ≤ 2
5. Myelosuppressive chemotherapy naive
6. Scheduled to receive and anticipated to complete the following chemotherapy regimen

   1. FEC (fluorouracil/epirubicin (100) / cyclophosphamide) (3 cycles);
   2. Docetaxel (3 cycles) chemotherapy
7. White blood cells (WBC) ≥ 3 × 10^9/L; Absolute neutrophil count (ANC) ≥ 2.0 × 10^9/L; platelet count ≥ 100 × 10^9/L; and hemoglobin ≥ 10 g/dL (6.2 mmol/L)
8. Adequate cardiac function (e.g. LVEF > 50% as determined by standard care) and adequate hepatic function (e.g. liver transaminases < 2.5 x ULN)
9. Women of childbearing potential with a negative serum pregnancy test and using a highly effective method of birth control (i.e. one that results in a less than 1% per year failure rate when used consistently and correctly, such as implants, injectables, combined oral contraceptives and intrauterine devices (IUDs)). Periodic abstinence is not an acceptable contraceptive method during the study period.

Exclusion Criteria: A subject will not be enrolled if any they meet any of the following criteria:

1. Known hypersensitivity to E.coli derived products or polyethylene glycol
2. No other malignancy except carcinoma in situ and basal-cell and squamous cell carcinoma of the skin, unless the other malignancy was treated ≥ 5 years ago with curative intent
3. Evidence of myelodysplasia, aplastic anemia, myelofibrosis, rheumatoid arthritis, systemic lupus erythematosus, or sickle cell disease
4. Clinical diagnosis or history of chronic infection such as hepatitis B virus (HBV), hepatitis C virus (HCV) or Human immunodeficiency virus (HIV) or history of tuberculosis
5. Previous exposure to filgrastim, perfilgrastim or lipegfilgrastim within 30 days before randomization
6. Treatment with systemically active antibiotics within 72 hours before chemotherapy
7. Chronic use of oral corticosteroids
8. Participation in a pharmacological clinical trial within 30 days before randomization
9. Clinical diagnosis of drug abuse or substance abuse within 30 days prior to screening
10. Documented alcohol abuse within 30 days prior to screening
11. Unwilling and/or not capable of ensuring compliance with the provisions of the study protocol
12. Pregnant or breastfeeding women where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive serum HCG laboratory test
13. Other serious medical condition that would prevent individual from receiving protocol treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 9 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-05-22 (Actual)

PRIMARY OUTCOMES:
Duration of neutropenia grade 1 or worse (absolute neutrophil count [ANC] ≤ 2.0 x 10^9/L) in the first cycle of chemotherapy (FE100C). | 21 days

SECONDARY OUTCOMES:
Duration of neutropenia grade 1 or worse (absolute neutrophil count [ANC] ≤ 2.0 x 10^9/L) in the fourth cycle of chemotherapy (docetaxel). | 21 days
Duration of severe neutropenia (ANC < 0.5 x 10^9/L) during the first chemotherapy cycle (21-day cycle FE100C) | 21 days
Duration of severe neutropenia (ANC < 0.5 x 10^9/L) during the fourth chemotherapy cycle (21-day cycle docetaxel) | 21 days
Incidence of severe neutropenia (ANC < 0.5 x 10^9/L) during all chemotherapy cycles | ~ 128 ± 2 days
Incidence and duration of febrile neutropenia defined as peak temperature ≥38.5°C and ANC < 0.5 x 10^9/L, during all chemotherapy cycles | ~ 128 ± 2 days
Incidence and duration of febrile neutropenia defined as peak temperature ≥38.0°C for two readings over two hours and ANC < 0.5 x 10^9/L, during all chemotherapy cycles | ~ 128 ± 2 days
Incidence and duration of infection and infection-related events based on use of antibiotics during all chemotherapy cycles | ~ 128 ± 2 days
Incidence and duration of infection and infection-related events based on the need for hospitalization during all chemotherapy cycles | ~ 128 ± 2 days
Incidence and duration of moderate (ANC ≥ 50 x 10^9/L) leukocytosis during all chemotherapy cycles | ~ 128 ± 2 days
Incidence and duration of severe (ANC ≥ 100 x 10^9/L) leukocytosis during all chemotherapy cycles | ~ 128 ± 2 days
Clinically meaningful changes in vital signs during all chemotherapy cycles - Assessment of Blood pressure | ~ 128 ± 2 days
  Assessment of Blood pressure (systolic and diastolic) helps determine the safety of the medications under study - ANF-RHO and Neulasta
Clinically meaningful changes in vital signs during all chemotherapy cycles - Assessment of Heart rate | ~ 128 ± 2 days
  Assessment of Heart rate helps determine the safety of the medications under study - ANF-RHO and Neulasta
Clinically meaningful changes in vital signs during all chemotherapy cycles - Assessment of Respiratory rate | ~ 128 ± 2 days
  Assessment of Respiratory rate helps determine the safety of the medications under study - ANF-RHO and Neulasta
Clinically meaningful changes in vital signs during all chemotherapy cycles - Assessment of Body Temperature | ~ 128 ± 2 days
  Assessment of Respiratory rate helps determine the safety of the medications under study - ANF-RHO and Neulasta
Incidence of bone pain, determined by a numerical rating scale, as well as other reported adverse events | ~ 128 ± 2 days
Duration of bone pain, determined by a numerical rating scale, as well as other reported adverse events | ~ 128 ± 2 days
Severity of bone pain, determined by a numerical rating scale, as well as other reported adverse events | ~ 128 ± 2 days
Site of bone pain, determined by a numerical rating scale, as well as other reported adverse events | ~ 128 ± 2 days
Pharmacokinetic profile of ANF-RHO and Neulasta - Measurement of Maximum Plasma Concentration (Cmax) | ~ 128 ± 2 days
  Cmax is the maximum concentration of the drug (either ANF-RHO or Neulasta) that is achieved after administration of a dose
Pharmacokinetic profile of ANF-RHO and Neulasta - Measurement of Time taken to reach the maximum concentration (Tmax) | ~ 128 ± 2 days
  Tmax is the time taken to reach the maximum concentration (Cmax) after administration of a dose.
Pharmacokinetic profile of ANF-RHO and Neulasta - Measurement of half-life (T1/2) | ~ 128 ± 2 days
  T1/2 is the time taken for ANF-RHO and Neulasta to reach half the value of their initial concentrations. T1/2 determination helps in understanding the duration for which ANF-RHO or Neulasta would be active upon administration.
Pharmacokinetic profile of ANF-RHO and Neulasta - Area Under the Curve (AUC[0-t]) | ~ 128 ± 2 days
  AUC[0-t] is an important parameter for determining as to how much of the drug is available in the body after administration of a drug formulation, in this case ANF-RHO vs Neulasta. Understanding the AUC for both these drug formulations will help us to determine the efficacy and safety profiles of these medicines.
Pharmacokinetic profile of ANF-RHO and Neulasta - Area Under the Curve (AUC[0-∞]) | ~ 128 ± 2 days
  Similar to AUC[0-t] which is estimated till time 't', in AUC[0-∞], the estimation is done on the concentration of the drug to an infinite time. Calculation of the AUC[0-∞], helps understand how much of the drug is available in the body at extremely low concentrations, beyond the limits of measurable concentrations.
Pharmacokinetic profile of ANF-RHO and Neulasta - Area Under the Curve (AUC[0-t]/AUC[0-∞]) | ~ 128 ± 2 days
  The parameter AUC[0-t]/AUC[0-∞] is useful to calculate the fraction of the Total AUC that was added due to the extrapolated AUC (AUC[0-∞]). It helps understand if the methods employed for determining the total AUC and drug's availability in the body are correct.
Incidence of anti-drug antibodies to ANF-RHO and Neulasta | ~ 128 ± 2 days

CONTACTS AND LOCATIONS:
Locations (8):
- France (4):
  - Hôpital Saint Louis - Center des Maladies du Sein, Paris
  - Institut de cancérologie Jean Godinot, Reims
  - Strasbourg Oncologie Libérale, Strasbourg
  - CHU de Tours, Tours
- Netherlands (4):
  - Erasmus Medical Center, Rotterdam
  - Ikazia Ziekenhuis, Rotterdam
  - Maasstad Ziekenhuis, Rotterdam
  - Franciscus Gasthuis & Vlietland, Schiedam

IPD SHARING:
Plan to Share IPD: No